CLINICAL TRIAL: NCT06837636
Title: The Use of Esophageal Pressure as a Guide to Set One Lung Ventilation During Capnothorax.
Brief Title: During Chest Surgery, One Lung is Isolated From Ventilation to Improve Visibility, With Carbon Dioxide Introduced Between the Lung and Chest Wall (Capnothorax): the Study Seeks to Optimize Ventilation Through Esophageal Pressure Measurement, Reducing Respiratory Complications.
Acronym: CapnoPes
Status: Not yet recruiting | Type: Observational
Sponsor: Cardarelli Hospital (Other)
Responsible Party: Principal Investigator, Gianluigi Lauro, Dr. Gianluigi Lauro,Anesthesiologist and critical care physician working in thoracic surgery and intensive care at Cardarelli Hospital, medical director., Cardarelli Hospital
Other Study IDs: 7029012025
Record Dates: First submitted 2025-02-15; First posted 2025-02-20 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Capnothorax; One Lung Ventilation; Thoracic Surgery; Esophageal Pressure Measurement
Keywords: capnothorax; one lung ventilation; esophageal pressure; thoracic surgery

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- CapnoPes

SUMMARY:
The objective of this single-center observational study is to improve the safety and effectiveness of chest surgery through the use of a new ventilation technique. During the operation, to allow the surgeon to work more precisely, only one lung will receive air from the respirator. To improve visibility during surgery, a small amount of carbon dioxide is introduced into the space between the lung and the chest wall, a procedure called capnothorax. The aim of the research is to find the best way to set the patient's ventilation during the operation, ensuring adequate oxygenation and minimizing the risks to the lung. To do this, we will use a method of measuring the pressure inside the esophagus, which will allow us to better understand the status of the lungs and adjust ventilation accordingly. Esophageal pressure is an indirect measure of the pressure within the lung. By measuring this pressure, we can get important information about the status of the lungs and their ability to expand and contract. By measuring esophageal pressure, researchers will be able to set ventilation more precisely, optimizing the amount of air that is supplied to the lungs and the pressure inside the lungs themselves. This could help prevent lung damage and improve the patient's breathing during and after surgery, reducing respiratory complications and improving patients' quality of life.

General data collected at the beginning of the study and before the surgical intervention:

* date of birth, gender, weight, and height,
* information and scores regarding the fitness for general anesthesia techniques,
* anesthesia risk assessment made by the American Society of Anesthesiologists (ASA),
* data related to respiratory mechanics.

Data collected during the surgical intervention:

* data related to respiratory mechanics measured at the ventilator,
* data recorded by the optivent monitor to which the esophageal probe is connected,
* hemodynamic data collected through a semi-invasive arterial blood pressure monitoring system,
* arterial blood gas analysis,
* pulmonary ultrasound findings.

DETAILED DESCRIPTION:
The aim of the study is to evaluate whether esophageal pressure can be useful in titration of adequate positive end-expiratory pressure (peep) during one-lung ventilation in robotic thoracic surgery, with repeated measurements on a single group of patients, to prevent atelectrauma, barotrauma, (VILI) ventilator-induced lung injury and post-operative pulmonary complications. The analysis will be carried out by analyzing the patients' medical records and data collection forms.

Study phase 1: screening for inclusion and informed consent, phase 2: monitoring and analysis of intraoperative data.

All patients will be subjected to general anesthesia with positioning of the double-lumen tube, with subsequent control of the correct positioning with the fiber bronchoscope. A volume-controlled ventilation mode will be set, so as to have an expiratory transpulmonary pressure (ptp exp) according to Talmor above 0 and a derived transpulmonary inspiratory pressure < 20 (according to Gattinoni) in each phase of ventilation. The Nutrivent tube is then positioned for the measurement of esophageal pressure and hemodynamic monitoring through semi-invasive blood pressure measurement. Then there is the positioning of the patient in lateral or semilateral decubitus and the OLV and after the capnothorax, the alveolar recruitment maneuver is carried out.

Measurements of ventilatory mechanics parameters and blood gas analysis will be carried out after:

* 15 minutes after induction of general anesthesia in two-lung ventilation (TLV) and in one lung ventilation (OLV),
* after positioning in lateral/semilateral decubitus in TLV and OLV,
* after capnothorax and alveolar recruitment maneuver in OLV,
* after 60 minutes from the ventilation set in OLV,
* every 60 minutes from the last recruitment step and/or alveolar recruitment maneuver in OLV,
* at the end of the capnothorax and in the supine position in TLV. After waking up, the LUS score (Lung Ultrasound) will be evaluated on the unoperated lung.

For the analysis of primary and secondary endpoints, appropriate descriptive and inferential statistical methodologies will be used. Continuous variables will be summarized using means and standard deviations in the case of normal distribution, while medians and interquartile ranges will be used for variables with non-normal distribution. Categorical variables will be described with absolute frequencies and percentages. This descriptive analysis will allow us to have a detailed picture of the characteristics of the population under study.

For the analysis of the primary endpoints, a repeated measures MANOVA will be used to evaluate the correlations between the P/F ratio, driving pressure and esophageal pressure during the different phases of OLV. This statistical approach is particularly suitable because it allows multiple related dependent variables to be analyzed simultaneously, providing a deeper understanding of the interactions between respiratory variables and esophageal pressure. The Greenhouse-Geisser correction will be applied if necessary to account for any violations of the sphericity assumption. The Greenhouse-Geisser correction will be applied if necessary to account for any violations of the sphericity assumption. According to the analysis performed with G*Power, an f test was used for a repeated measures MANOVA with a single group and four measurements. The effect size (f) was set at 0.30, with a significance level (α) of 0.05 and a desired statistical power of 0.90. The correlation between repeated measurements was taken to be 0.2 and the non-sphericity correction (ε) was set to 0.8. The results of the analysis indicated a noncentrality parameter (λ) of 16.20, with a critical f value of 2.89. The degrees of freedom of the numerator and denominator are 3.0 and 33.0, respectively. The total sample size required was found to be 36 participants, with an effective power of 0.904, which meets the intended goal of statistical power. Since the study involves only one group and the postoperative complications variable is binary (present/absent), the binomial test will be used to describe the proportion of patients who develop postoperative complications compared to a theoretical expected proportion of 20%, obtained from the literature. This test was chosen because it is suitable for small samples and allows for a significant statistical evaluation of postoperative complications without the need to correlate this variable with other categorical variables. This approach will provide an accurate overview of complications within the study population. A value of p < 0.05 will be considered statistically significant. Results will be reported as mean ± sd for continuous variables. Statistical analysis will be performed using Rstudio software (version 2023.09.0+351). Furthermore, the sample size calculation was performed with the G*Power software (version 3.1).

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years • Patients to undergo robotic thoracic surgery with capnothorax

Exclusion Criteria:

* Pre-existing cardiac and/or pulmonary pathologies resulting in an ASA > 3

  * Contraindications to the placement of a nasogastric tube
  * Severe COPD (stage 3 or 4)
  * Emergency thoracotomy or sternotomy for surgical complications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients from the AORN "Antonio Cardarelli" of Naples undergoing robotic thoracic surgery will be selected and will receive one-lung ventilation during general anesthesia with the capnothorax
Sampling Method: Non-Probability Sample
Enrollment: 36 (Estimated)
Dates: Start 2025-02-20 (Estimated); Primary Completion 2026-02-20 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Evaluate the P/F ratio (PaO2/ FiO2), the driving pressure during the OLV phases in relation to the esophageal pressure. | from induction of general anesthesia to awakening
  Evaluate the P/F ratio (PaO2/ FiO2) and the driving pressure (the difference between plateau pressure and PEEP, during the OLV phases in relation to the esophageal pressure.

SECONDARY OUTCOMES:
P/F upon awakening from general anesthesia and evaluate postoperative respiratory complications | within 24 hours post-operatively
  Evaluate the P/F upon awakening from general anesthesia and evaluate post-operative respiratory complications with the LUS score.The LUS (Lung Ultrasound Score) is a scoring system used to assess lung involvement. It is based on ultrasound images of the lungs, where different areas of the chest are evaluated for the presence of B-lines, consolidations, and other abnormalities. Each lung zone is scored, helping to classify the severity of the condition and monitor its clinical progression. This method is non-invasive and effective for real-time assessment.

CONTACTS AND LOCATIONS:
Locations (1):
- Azienda Ospedaliera di Rilievo Nazionale ed Alta Specializzazione "Antonio Cardarelli", Napoli, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cammarota G, Lauro G, Santangelo E, Sguazzotti I, Perucca R, Verdina F, Boniolo E, Tarquini R, Bignami E, Mongodi S, Arisi E, Orlando A, Della Corte F, Vaschetto R, Mojoli F. Mechanical Ventilation Guided by Uncalibrated Esophageal Pressure May Be Potentially Harmful. Anesthesiology. 2020 Jul;133(1):145-153. doi: 10.1097/ALN.0000000000003327. PMID 32349074
- [Background] Yoshida T, Amato MBP, Grieco DL, Chen L, Lima CAS, Roldan R, Morais CCA, Gomes S, Costa ELV, Cardoso PFG, Charbonney E, Richard JM, Brochard L, Kavanagh BP. Esophageal Manometry and Regional Transpulmonary Pressure in Lung Injury. Am J Respir Crit Care Med. 2018 Apr 15;197(8):1018-1026. doi: 10.1164/rccm.201709-1806OC. PMID 29323931
- [Background] Wang QY, Zhou Y, Wang MR, Jiao YY. Effects of starting one lung ventilation and applying individualized PEEP right after patients are placed in lateral decubitus position on intraoperative oxygenation for patients undergoing thoracoscopic pulmonary lobectomy: study protocol for a randomized controlled trial. Trials. 2024 Jul 22;25(1):500. doi: 10.1186/s13063-024-08347-8. PMID 39039591
- [Background] Gattinoni L, Chiumello D, Carlesso E, Valenza F. Bench-to-bedside review: chest wall elastance in acute lung injury/acute respiratory distress syndrome patients. Crit Care. 2004 Oct;8(5):350-5. doi: 10.1186/cc2854. Epub 2004 May 7. PMID 15469597
- [Background] Ferrando C, Carraminana A, Pineiro P, Mirabella L, Spadaro S, Librero J, Ramasco F, Scaramuzzo G, Cervantes O, Garutti I, Parera A, Argilaga M, Herranz G, Unzueta C, Vives M, Regi K, Costa-Reverte M, Sonsoles Leal M, Nieves-Alonso J, Garcia E, Rodriguez-Perez A, Farina R, Cabrera S, Guerra E, Gallego-Ligorit L, Herrero-Izquierdo A, Valles-Torres J, Ramos S, Lopez-Herrera D, De La Matta M, Gokhan S, Kucur E, Mugarra A, Soro M, Garcia L, Sastre JA, Aguirre P, Salazar CJ, Ramos MC, Morocho DR, Trespalacios R, Ezequiel-Fernandez F, Lamanna A, Pia Cantatore L, Laforgia D, Bellas S, Lopez C, Navarro-Ripoll R, Martinez S, Vallverdu J, Jacas A, Yepes-Temino MJ, Belda FJ, Tusman G, Suarez-Sipmann F, Villar J; iPROVE-OLV Research Network Group. Individualised, perioperative open-lung ventilation strategy during one-lung ventilation (iPROVE-OLV): a multicentre, randomised, controlled clinical trial. Lancet Respir Med. 2024 Mar;12(3):195-206. doi: 10.1016/S2213-2600(23)00346-6. Epub 2023 Dec 5. PMID 38065200
- [Background] Kiss T, Wittenstein J, Becker C, Birr K, Cinnella G, Cohen E, El Tahan MR, Falcao LF, Gregoretti C, Granell M, Hachenberg T, Hollmann MW, Jankovic R, Karzai W, Krassler J, Loop T, Licker MJ, Marczin N, Mills GH, Murrell MT, Neskovic V, Nisnevitch-Savarese Z, Pelosi P, Rossaint R, Schultz MJ, Neto AS, Severgnini P, Szegedi L, Vegh T, Voyagis G, Zhong J, de Abreu MG, Senturk M; PROTHOR investigators and the Research Workgroup PROtective VEntilation Network (PROVEnet) of the European Society of Anaesthesiology (ESA). Correction to: Protective ventilation with high versus low positive end-expiratory pressure during one-lung ventilation for thoracic surgery (PROTHOR): study protocol for a randomized controlled trial. Trials. 2019 May 8;20(1):259. doi: 10.1186/s13063-019-3371-y. PMID 31068212
- [Background] Yoon S, Nam JS, Blank RS, Ahn HJ, Park M, Kim H, Kim HJ, Choi H, Kang HU, Lee DK, Ahn J. Association of Mechanical Energy and Power with Postoperative Pulmonary Complications in Lung Resection Surgery: A Post Hoc Analysis of Randomized Clinical Trial Data. Anesthesiology. 2024 May 1;140(5):920-934. doi: 10.1097/ALN.0000000000004879. PMID 38109657
- [Background] Cammarota G, Lauro G, Sguazzotti I, Mariano I, Perucca R, Messina A, Zanoni M, Garofalo E, Bruni A, Della Corte F, Navalesi P, Bignami E, Vaschetto R, Mojoli F. Esophageal Pressure Versus Gas Exchange to Set PEEP During Intraoperative Ventilation. Respir Care. 2020 May;65(5):625-635. doi: 10.4187/respcare.07238. PMID 32345760
- [Background] Peel JK, Funk DJ, Slinger P, Srinathan S, Kidane B. Positive end-expiratory pressure and recruitment maneuvers during one-lung ventilation: A systematic review and meta-analysis. J Thorac Cardiovasc Surg. 2020 Oct;160(4):1112-1122.e3. doi: 10.1016/j.jtcvs.2020.02.077. Epub 2020 Feb 29. PMID 32276803
- [Background] Reinius H, Borges JB, Engstrom J, Ahlgren O, Lennmyr F, Larsson A, Freden F. Optimal PEEP during one-lung ventilation with capnothorax: An experimental study. Acta Anaesthesiol Scand. 2019 Feb;63(2):222-231. doi: 10.1111/aas.13247. Epub 2018 Aug 21. PMID 30132806